CLINICAL TRIAL: NCT05478122
Title: Soft Mist Spray Device for Airway Anaesthesia During Awake Videolaryngoscopy
Acronym: CT2Trachospray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT2 Trachospray
Record Dates: First submitted 2022-07-25; First posted 2022-07-28 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-07

CONDITIONS: Airway; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Subjects will be asked to inhale 4 ml lidocaine 4% via the Trachospray device
  Interventions: Device: Trachospray for awake videolaryngoscopy

INTERVENTIONS:
Device: Trachospray for awake videolaryngoscopy — Subjects will be asked to inhale 4 ml lidocaine 4% via the Trachospray device

SUMMARY:
Rationale:

Effective and fast topical anaesthesia of the upper airway is of paramount importance in awake (conscious) videolaryngoscopy of the airway in order to avoid patient discomfort. Different methods of anesthetizing the airway have been described. Conventional topical airway anaesthesia is not always effective due to non-optimal flow patterns and generation of ineffective local anaesthetic aerosols. Other methods of anaesthetizing the airway are more invasive. In order to optimize topical anaesthesia of the airway a soft mist spray device (Trachospray) for topical anaesthesia of the airway has been developed, in which optimal airflow patterns are obtained and local anaesthetic aerosols are generated which will reach the target zone for anesthetizing the airway.

Objective: In this study, the Trachospray will be used for awake videolaryngoscopy, to evaluate its use, effectiveness and comfort level for patients and anaesthesiologist.

Study design: Interventional study.

Study population: 20 healthy human volunteers, ASA 1, 18-60 years old.

Intervention: Subjects will be asked to inhale 4 ml lidocaine 4% via the Trachospray device

Main study parameters/endpoints:

Anaesthesia of the airway as evaluated with successful awake videolaryngoscopy with minimal discomfort for the subject.

Nature and extent of the burden and risks associated with participation:

Risk management on the Trachospray device shows that all user risks are mitigated and no residual risks remain for the use of the device. Testing of the device and the application of the device in daily practice has no additional risks than the present technique of performing anaesthesia of the airways.There may be some discomfort during the procedure, mainly airway irritation which may cause coughing or gag reflex.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-60 years
* Lean body weight >= 50 kg
* ASA physical status 1

Exclusion Criteria:

* Inability to cooperate with adequate airway assessment,
* History of hepatic, renal and coagulation diseases,
* Respiratory tract pathology
* Pregnancy
* Risk of regurgitation or aspiration
* Allergy to amide type of local anaesthetics
* No written informed consent by subject

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
Complete anaesthesia of the airway as evaluated with successful awake videolaryngoscopy with minimal discomfort for the subject | 3 months
  Discomfort and level of anesthesia will be measured with a numerical rating scale (NRS). 60 / 5.000 Vertaalresultaten So the result will be displayed in whole numbers.

CONTACTS AND LOCATIONS:
Overall Officials: Geert-Jan van Geffen, Principal Investigator — Radboud University Medical Center (Radboudumc); Hielke Markerink, Study Director — Radboud University Medical Center (Radboudumc); Jorgen Bruhn, Study Chair — Radboud University Medical Center (Radboudumc)
Locations (1):
- Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No